CLINICAL TRIAL: NCT04938492
Title: The Association Between Loneliness and Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lisham Ashrafioun, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005387
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Opioid Use; Loneliness
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (CBT) (Experimental): CBT delivered over the course of 6, ~45 minute sessions delivered via telehealth.
  Interventions: Behavioral: Cognitive Behavioral Therapy for loneliness (CBT-L)
- Health Education (Active Comparator): Health education sessions delivered over the course of 6, ~45 minute sessions delivered via telehealth.
  Interventions: Behavioral: Physical Health Education Training (PHET)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for loneliness (CBT-L) — 6 sessions focused on addressing thoughts, emotions, and behaviors that maintain feeling alone as a way to reduce loneliness and substance use.
  Arms: Cognitive Behavioral Therapy (CBT)
Behavioral: Physical Health Education Training (PHET) — Health education provides information on the importance and benefits of and guidelines for living a healthy lifestyle.
  Arms: Health Education

SUMMARY:
The proposed study will determine if cognitive behavioral therapy will help improve loneliness in people who use opioids.

DETAILED DESCRIPTION:
The proposed study will be the first to assess the cognitive, affective, and behavioral pathways by which loneliness impacts opioid use. Individuals with an opioid use disorder (OUD) reporting loneliness will be randomized to either a 6-session Cognitive- Behavioral Therapy for loneliness (CBT-L) or a 6-session education control condition, both delivered via telehealth. Telehealth delivery can be easily implemented and can increase reach and access to individuals not engaged in treatment. We will use an established brief CBT manual to address loneliness. We will assess loneliness, negative affect (i.e., depression and anxiety), and the quality and quantity of social interactions prior to, during, and after the intervention to evaluate the subsequent impact on opioid use trajectories. Participant will complete questionnaires pre-treatment, post-treatment, and at 1- and 2-months posttreatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be ages 18+
* Understand English
* Have internet access
* Screen positive for an active OUD on the OUD Module of the Structured Clinical Interview for DSM-5 (Diagnostic & Statistical Manual of Mental Disorder, 5th edition) Research Version (SCID-5-RV)
* Screen positive for loneliness by scoring at least a T-score > 60 on the NIH Toolbox Loneliness Scale

Exclusion Criteria:

* Consistent with previously used telehealth-delivered assessments, we will exclude any participant with cognitive impairment as measured by the Blessed Orientation-Memory-Concentration Test (BOMC)
* Potential participants who are in the process of detoxifying as measured by the Subjective Opiate Withdrawal Scale will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data is available upon request as part of scientific collaboration.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited from social networking platforms. Recruitment started 08/2021.
Pre-assignment Details: Participants in both conditions receive a baseline assessment and then are randomized to either CBT or Health Education.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy (CBT) | Health Education
Started | 63 | 62
Completed | 46 | 44
Not Completed | 17 | 18
Not completed — Lost to Follow-up | 17 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy (CBT) | Health Education | Total
Number analyzed (Participants) | 63 | 62 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.8) | 42.2 (9.7) | 43.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 27 | 26 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 58 | 58 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 19 | 32
  White | 45 | 39 | 84
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
UCLA Loneliness Scale [Mean (Standard Deviation); unit: units on a scale - loneliness] — Loneliness will be measured using the UCLA Loneliness Scale. A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as 1 (never), 2 (rarely), 3 (sometimes) or 4 (often). The scores range from 20-80 with higher scores indicating worse outcome.
  units on a scale - loneliness | 58.0 (9.1) | 58.5 (7.9) | 58.2 (8.5)
Duke Social Support Index-Perceived Social Support [Mean (Standard Deviation); unit: units on a scale] — Duke Social Support Index-Perceived Social Support subscale assesses perceived social support. Higher scores indicate a higher perceived social support. Scores range from 6 to 18.
  units on a scale | 11.4 (2.9) | 11.7 (3.1) | 11.5 (3.0)
Percent days abstinent from opioids [Mean (Standard Deviation); unit: percentage of days] — Participants will complete a calendar indicating the type and frequency of drug use. Percent days abstinent from opioids is calculated by the number of days in which opioids were not used divided by the number of days in the assessment (i.e., 60).
  percentage of days | 40.7 (36.6) | 33.0 (34.6) | 36.9 (35.7)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Loneliness
Description: Loneliness will be measured using the University of California-Los Angeles (UCLA) Loneliness Scale. A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as 1 (never), 2 (rarely), 3 (sometimes) or 4 (often). The scores range from 20-80 with higher scores indicating worse outcome.
Time Frame: baseline to 2 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy (CBT) | Health Education
Number analyzed (Participants) | 46 | 44
score on a scale | -8.3 (14.9) | -10.3 (12.5)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy (CBT) vs Health Education; Test type: Superiority; p > .05, Latent growth modeling; Slope = 2.08

2. Secondary Outcome: Mean Change in Percent Days Abstinent From Opioids
Description: Participants will complete a calendar indicating the type and frequency of drug use.
Time Frame: baseline to 2 months post-treatment
Measure: Mean (Standard Deviation); unit: percentage of days (abstinent/total)
Arm/Group | Cognitive Behavioral Therapy (CBT) | Health Education
Number analyzed (Participants) | 46 | 44
percentage of days (abstinent/total) | 40 (43) | 20 (30)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy (CBT) vs Health Education; Test type: Superiority; p < .001, Latent growth modeling; Slope = .19

3. Secondary Outcome: Mean Change in Percent Days Abstinent From Other Drugs
Description: Participants will complete a calendar indicating the type and frequency of drug use.
Time Frame: baseline to 2 months
Measure: Mean (Standard Deviation); unit: percentage of days (abstinent/total)
Arm/Group | Cognitive Behavioral Therapy (CBT) | Health Education
Number analyzed (Participants) | 46 | 44
percentage of days (abstinent/total) | 30 (42) | 14 (33)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy (CBT) vs Health Education; Test type: Superiority; p < .01, Latent growth modeling; Slope = .22

4. Secondary Outcome: Mean Change in Social Support
Description: Duke Social Support Index assesses several domains of perceived social support, including social network size, social interaction, social satisfaction, and instrumental social support. Higher scores indicate a higher quality of social interactions or perceived social support. Scores range from 6 to 18.
Time Frame: baseline to 2 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy (CBT) | Health Education
Number analyzed (Participants) | 46 | 44
score on a scale | 1.6 (3.4) | 1.0 (3.0)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy (CBT) vs Health Education; Test type: Superiority; p > .05, Latent growth modeling; Slope = .23

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of approximately 4 months from baseline to 2-months post-treatment.
Arm/Group | Cognitive Behavioral Therapy (CBT) | Health Education
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 1/63 | 1/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (CBT) (N=63) | Health Education (N=62)
increase in psychiatric distress (Psychiatric disorders) | 1 (1) | 0 (0)
drug withdrawal (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT04938492/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT04938492/ICF_000.pdf